CLINICAL TRIAL: NCT03788642
Title: Efficacy of Low-level Laser Therapy for the Treatment of Diabetic Foot Ulcer
Brief Title: Low-level Laser Therapy for the Treatment of Diabetic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Si475/2561
Record Dates: First submitted 2018-12-25; First posted 2018-12-27 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer; Low Level Laser Therapy
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Intervention Model Description: The randomised clinical trial with participants randomised1:1 to either
  * Control group : Patients will wear LED shoe (Placebo) 30 minutes once daily
  * Laser group : Patients will wear Laser shoe 30 minutes once daily
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control LED Shoe arm (Active Comparator): Patients with DFU will wear LED shoe 30 minutes per day
  Interventions: Procedure: Control LED shoe arm
- Laser Shoe arm (Active Comparator): Patients with DFU will wear Laser shoe 30 minutes per day
  Interventions: Procedure: Laser Shoe arm

INTERVENTIONS:
Procedure: Control LED shoe arm — Patients with DFU will wear LED shoe 30 minutes once daily
  Arms: Control LED Shoe arm
Procedure: Laser Shoe arm — Patients with DFU will wear Laser shoe 30 minutes once daily
  Arms: Laser Shoe arm

SUMMARY:
The study evaluates the efficacy of Low-level laser therapy on ulcer healing in patients with diabetic foot ulcer. Half the patients are randomized to receive Low-level laser therapy and a half to recieve the placebo (LED).

DETAILED DESCRIPTION:
Low-level laser therapy(LLLT) has been reported to aid ulcer healing in patients with diabetic foot ulcer. However, patients need to come to hospital to receive LLLT performed by medical professional. The LLLT shoe has been developed for home using. Patients can wear LLLT shoe 30 min once daily instead of going hospital for LLT therapy. The aim of this study is to see whether LLLT shoe helps with healing compare with placebo (LED shoe).

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic diabetic foot ulcer
* Ankle brachial index ≥ 0.4
* Toe pressure brachial index ≥ 0.3
* Transcutaneous oxygen measurement (TCOM) ≥ 40 mmHg
* Ulcer size less than 25 cm2

Exclusion Criteria:

* Infected ulcer
* Fever
* HbA1C > 15 %

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Ulcer Healing Rate | 12 weeks
  Healing rate of control and laser group will be reported at 12 weeks

SECONDARY OUTCOMES:
Time to ulcer healing | time from date of randomisation to date of healing within the 12 month study period
  For the purposes of this study, ulcer healing is defined as complete re-epithelialization of all ulceration on the randomized leg in the absence of a scab (eschar) with no dressing required.
Clinical Success - Complications | up to 12 months
  Incidence of complications related to the LLT shoe

CONTACTS AND LOCATIONS:
Overall Officials: Nuttawut SERMSATHANASAWADI, MD, PhD, Principal Investigator — Mahidol University
Locations (1):
- Vascular Surgery, Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand